CLINICAL TRIAL: NCT06412133
Title: Conversations in Light and Shadow: Assessing Phototherapy's Impact on Breast Cancer Patients: Study Protocol for a Multicenter, Randomized Controlled Trial
Brief Title: Conversations in Light and Shadow: Assessing Phototherapy's Impact on Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yun-Chen Chang (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Sponsor-Investigator, Yun-Chen Chang, assistant professor, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CMUH113
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Breast Cancer Female; Randomized Controlled Trial
MeSH Terms: conditions — Breast Neoplasms | interventions — Photography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): photography therapy
  Interventions: Behavioral: photography

INTERVENTIONS:
Behavioral: photography — This study examines the impact of phototherapy intervention on anxiety, stress, and body image among breast cancer patients. Participants engaged in a five-week, one-on-one session series, utilizing a pre-post-test design with parallel groups.

SUMMARY:
This study examines the impact of phototherapy intervention on anxiety, stress, and body image among breast cancer patients. Participants engaged in a five-week, one-on-one session series, utilizing a pre-post-test design with parallel groups. Quantitative data were collected using the Depression Anxiety Stress Scales (DASS-21) and the Body Image Scale. In addition to quantitative measures, in-depth individual interviews were conducted to gather qualitative data. The combined data were then analysed to assess the effectiveness of the intervention.

DETAILED DESCRIPTION:
Background: Breast cancer ranks as the most prevalent cancer among women in Taiwan. According to statistical data, breast cancer patients face a risk of recurrence ranging from 4.7% to 50% within five years' post-treatment. The repeated cycles of occurrence and treatment not only cause physiological changes but also significant psychological stress, particularly in response to mastectomies and altered body image perceptions, all of which can adversely affect quality of life. However, current interventions in Taiwan, such as phototherapy, primarily aim to improve life quality and intimate relationships, with scant in-depth research focusing on the impacts on body image.

Objective: This study investigates whether phototherapy intervention can ameliorate psychological issues in breast cancer patients by focusing on three aspects: anxiety, stress, and body image. The research aims to address gaps in existing knowledge regarding the effectiveness of such interventions on these specific psychological dimensions.

Design and Methods: This study examines the impact of phototherapy intervention on anxiety, stress, and body image among breast cancer patients. Participants engaged in a five-week, one-on-one session series, utilizing a pre-post-test design with parallel groups. Quantitative data were collected using the Depression Anxiety Stress Scales (DASS-21) and the Body Image Scale. In addition to quantitative measures, in-depth individual interviews were conducted to gather qualitative data. The combined data were then analysed to assess the effectiveness of the intervention.

Setting(s): The study will be conducted across five medical centers in Taiwan.

Participants: The study included 1-3 stage breast cancer patients aged between 20 and 55 years who provided informed consent. Due to the exploratory nature of the research, a formal sample size analysis was not conducted. However, it was deemed that the anticipated sample size for the quantitative aspect of the study was sufficiently large (n =78) to obtain precise point estimates. Interventions were planned to be allocated to eligible breast cancer patients in a 1:1 ratio. Variables will be described using absolute and relative frequencies, means, medians, and relevant distribution estimates based on the measurement level. The primary outcomes will be described using paired t-tests and independent-samples t-tests.

Results: The study commenced in September 2024, with results expected to be available by July 2025.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage 1-3 breast cancer within the past five years,
* Aged between 20 and 55 years,
* Ability to communicate in Mandarin or Taiwanese,
* Ownership of a mobile phone and proficiency in using it for photography,
* Willingness to participate in the study, and capacity to provide informed consent

Exclusion Criteria:

* Individuals with a documented history of severe mental illness,
* Diagnosis of stage 4 breast cancer
* Current engagement in other adjunctive therapies

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-09-17 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | 5 weeks
  Depression Anxiety Stress Scales (DASS-21) developed by Lovibond and Lovibond (1995) is a structured emotional assessment tool. Higher scores on the scale indicate higher levels of depression, anxiety, and stress. The Cronbach's α values for the depression, anxiety, and stress subscales are 0.94, 0.87, and 0.91, respectively, indicating good reliability and internal consistency. The current prevalent version consists of 21 items (DASS-21), with scores interpreted as follows: 0 means "does not apply to me at all," 1 means "applies to me to some degree, or some of the time," 2 means "applies to me to a considerable degree, or a good part of the time," and 3 means "applies to me very much, or most of the time."
body image scale (BIS) | 5 weeks
  Body Image Scale used in this study was assessed by Hopwood et al. (2001) among breast cancer patients, with an internal consistency Cronbach's α value of 0.85. After re-assessment among breast cancer patients, the internal consistency Cronbach's α value improved to 0.93, indicating good reliability and test-retest reliability. This study utilized the Body Image Scale translated by Lin (2009) for assessment. This scale consists of 10 reverse-scored questions, with scores ranging from 10 to 40. Higher scores indicate a more negative body image tendency.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung, Beitun Dist
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No